CLINICAL TRIAL: NCT06408701
Title: Modeling Ocular Developmental Diseases From 3D Cultures of Optic Vesicle Organoids Derived From hiPSCs of Patients With Ocular Malformations
Acronym: OrganoEye
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0626
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Eye Abnormalities
Keywords: Microphthalmia; Anophthalmia; Coloboma; Aniridia
MeSH Terms: conditions — Eye Abnormalities; Microphthalmos; Anophthalmos; Coloboma; Aniridia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects presenting with an ocular developmental anomaly: Biological samples will be collected in the normal diagnosis and follow-up process
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Blood will be taken in larger quantity

SUMMARY:
Ocular morphogenesis is a complex process starting as early as the 4th week of embryonic life, involving interactions between varioustissues of different origin and conserved genes. Anomalies in ocular development , often of genetic origin, pose diagnostic and therapeutic challenges. Animal models are limited, so human-induced pluripotent stem cell (hiPSC)-derived optic vesicle containing brain organoids (OVBOs) offer a promising alternative. These pathological OVBOs, created from patients' cells with ocular malformations, allow for the study of underlying molecular mechanisms and testing of therapies.

DETAILED DESCRIPTION:
The eye's ability to perform its visual functions depends on its three-dimensional structure. Ocular morphogenesis is a complex process that begins in humans as early as the 4th week of embryonic life, requiring coordinated interactions between various embryologically diverse tissues involving highly conserved genes (Cardozo MJ, 2023). Disruption in any of these stages of ocular development, due to genetic, toxic, or environmental factors, can result in growth or formation defects of the eye globe. Among the most frequent ocular developmental anomalies , there are micro-anophthalmia, coloboma, anterior segment dysgenesis and aniridia (Plaisancie J, 2019). Most of these anomalies are of genetic origin. The primary obstacle in understanding these diseases is the lack of easily accessible tissue for sampling, which would allow for expression analyses and the study of underlying molecular mechanisms.

In this group of pathologies, understanding the pathophysiological mechanisms and therapeutic development was until recently quite limited and relied almost exclusively on the establishment of genetically modified animal models, a procedure that is lengthy, costly, and cumbersome. Moreover, routine diagnostic use of this model is not feasible in a hospital setting. Therefore, it is necessary to develop new tools and models to advance the understanding and management of these pathologies. The use of human induced pluripotent stem cells (hiPSCs) now allows for the understanding of the complexity of early organ development through the generation of 3D cellular models. Indeed, recent studies have shown that hiPSC-derived brain organoids retain, in a specific culture environment, the intrinsic capacity to develop optic vesicles (OV) mimicking early physiological ocular development and containing various ocular tissues (Gabriel E, 2021).

The optic vesicle organoid (OVBO) model thus represents a preferred alternative to the animal model in studying pathophysiological mechanisms and their use in preclinical trials. In addition to ethical and financial considerations, the latter has numerous advantages, particularly allowing the study of defective mechanisms directly from patient cells (precision medicine). Researchers have already developed the OVBO model from control hiPSC lines and have characterized the model under "physiological" conditions.

The next step in understanding the model and proving its utility in patients relies on studying the induced phenotype in OVBO models generated from hiPSCs from patients with genetically characterized ocular malformations. These "pathological" OVBO models will allow for detailed study of the molecular and cellular bases involved in these patients. Once the relevance of the model is demonstrated in modeling developmental pathologies of the eye, researchers will attempt to show that the OVBO model constitutes a robust alternative to the murine model in preclinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated with a social security scheme.
* Patients with ocular malformations.
* Signed informed consent obtained from the patient and/or their legal representatives.

Exclusion Criteria:

* Inability to understand the nature and objectives of the study and/or difficulties in communicating with the investigator.
* Deprivation of liberty by judicial or administrative decision.
* Any other pathological or psychological condition deemed incompatible by the investigator for the proper conduct of the study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: These patients will be solicited/sampled based on the genetic origin of the malformation they carry.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-05-02 (Estimated); Primary Completion 2034-05-02 (Estimated); Study Completion 2034-05-02 (Estimated)

PRIMARY OUTCOMES:
Culture of Optic Vesicles containing Brain Organoids (OVBOs) for the Study of Eye malformations | Day 60 of Development
  Macroscopic Examination and Expression of Specific Tissue Markers to Identify Optic Vesicle Anomalies

SECONDARY OUTCOMES:
Molecular and Cellular Study of Genetically Characterized Ocular Malformations in Patients | through study completion, an average of 1 year
  Identification of Genetic Basis for Observed Patient Pathology

CONTACTS AND LOCATIONS:
Overall Officials: Julie Plaisancie, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Purpan University Hospital, Toulouse, France